CLINICAL TRIAL: NCT03484143
Title: Vielight Neuro RX Gamma Photobiomodulation Device for Moderate to Severe Alzheimer's Disease
Brief Title: Neuro RX Gamma - Pivotal Phase
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been too slow. We are considering some changes to the protocol.
Sponsor: Vielight Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P17.03
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease
Keywords: Moderate to Severe Alzheimer's Disease,
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Neuro RX Gamma device (Active Comparator): Neuro RX Gamma device delivers low-energy near-infrared light, through 5 diodes, to the brain transcranially and intranasally
  Interventions: Device: Active Neuro RX Gamma device
- Sham Neuro RX Gamma device (Sham Comparator): Sham Neuro RX Gamma device is identical in appearance and sound as the active Neuro RX Gamma device but does not emit low-energy near infrared light
  Interventions: Device: Sham Neuro RX Gamma device

INTERVENTIONS:
Device: Active Neuro RX Gamma device — Twenty minute treatment session, 6 days a week for 24 weeks
  Arms: Active Neuro RX Gamma device
Device: Sham Neuro RX Gamma device — Twenty minute treatment session, 6 days a week for 24 weeks
  Arms: Sham Neuro RX Gamma device

SUMMARY:
The active Neuro RX Gamma device uses non-invasive near-infrared energy delivered to the brain with the intention to improve cognitive functioning and quality of life in patients with moderate to severe Alzheimer's Disease. Treatment will occur at home-based treatment sessions with the device.

DETAILED DESCRIPTION:
A potential participant will undergo pre-screening and screening assessments to assess eligibility for the study. Eligible participants will undergo a baseline visit in which they will be randomized to either active or sham Neuro RX Gamma device.

The Vielight Neuro RX Gamma is a non-invasive device that administers low-energy near-infrared LED (light emitting diode) light to the brain transcranially and intranasally.

There are two treatment phases in the trial, each with a duration of 12 weeks. The patient along with the caregiver will perform home (or living facility) - based treatments with the device and document the sessions in a patient diary. The device will be applied to the patient participant by a dedicated caregiver for a 20 minute daily session, 6 days a week for a total of 12 weeks. The study participant and caregiver will be required to return to the clinic for follow-up assessments at 12 and 24 weeks post randomization, between treatment phases.

228 patients will be enrolled across 12 sites in Canada and the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AD, defined as probable Alzheimer's disease of the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association.
2. Mini-mental state examination (MMSE) score between 8-20.
3. If receiving AD/psychotropic medication, must be on a stable dosage for at least 12 weeks prior to trial enrolment with no anticipated changes for the duration of the trial
4. Age 50 and older at the time of enrolment.
5. Severe Impairment Battery score at baseline ≤90
6. Adequate caregiver to ensure compliance of home-based treatments and to complete study assessments and questionnaires.

Exclusion Criteria:

1. Evidence of a relevant abnormality other than Alzheimer's disease on MRI or CT scan obtained within previous 24 months of enrolment into the trial, as listed below:

   1. Detection of more than 2 subcortical lacunar infarcts
   2. Any hemorrhage or infarct in a strategic location, such as the anterior nuclei of the thalamus (including dorso-medial nucleus)
   3. Space-occupying lesions compressing or compromising brain structures. (Note small meningiomas not compressing brain areas may be allowed)
   4. Patients with imaging findings that in the opinion of the investigator could be contributing to cognitive impairment (such as major cortical strokes, extensive white matter disease, etc.)

   Any patient without a scan in the past 2 years should undergo an MRI or CT as part of the study's screening assessment.
2. History of significant agitation and/or aggression.
3. History of stroke or epileptic seizures.
4. Current neurologic disease affecting cognition other than Alzheimer's disease.
5. Photosensitivity reactions to sunlight or visible light (polymorphous light eruption, solar urticaria, persistent light reactivity).
6. History of recurrent epistaxis within the last 24 weeks or currently taking major anti-coagulants (including warfarin, low molecular weight heparin)
7. Increased skin sensitivity at the treatment site including active herpes simplex in the treatment area, history of keloid formation, or history of retinoid use in the past month.
8. Pregnant or lactating or planning to become pregnant.
9. Currently undergoing light therapy treatment.
10. Current participation in another interventional clinical trial.
11. Any reason that, in the opinion of the investigator, might place a participant at unacceptable risk for participation in the trial.
12. Subject and/or caregiver does not speak English at a level necessary for the completion of the assessments.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in Severe Impairment Battery (SIB) score | Baseline to Week 24
  The SIB assesses cognitive abilities in severely impaired individuals. The scale covers social interaction, memory, orientation, language, attention, praxis, visuospatial ability, construction and orientation to name. There are 40 items with a total score range from 0-100. Scores of less than 63 on the SIB are rated as very severely impaired.
Change in Alzheimer's Disease Cooperative Study Activities of Daily Living for Severe Alzheimer's Disease (ADCS-ADL-Sev) | Baseline to Week 24
  The ADCS-ADL-Sev assesses the ability of patients with moderate to severe dementia to perform activities of daily living. There are 19 items with a total score range of 0-54.

SECONDARY OUTCOMES:
Change in Severe Impairment Battery (SIB) score | Baseline to Week 12
  The SIB assesses cognitive abilities in severely impaired individuals. The scale covers social interaction, memory, orientation, language, attention, praxis, visuospatial ability, construction and orientation to name. There are 40 items with a total score range from 0-100. Scores of less than 63 on the SIB are rated as very severely impaired.
Change in Alzheimer's Disease Cooperative Study Activities of Daily Living for Severe Alzheimer's Disease (ADCS-ADL-Sev) | Baseline to Week 12
  The ADCS-ADL-Sev assesses the ability of patients with moderate to severe dementia to perform activities of daily living. There are 19 items with a total score range of 0-54.
Change in European Quality of Life Scale (EQ-5 dimensions [5D], proxy version) | Baseline to Week 12 and Baseline to Week 24
  The EQ-5D is a standardized instrument for use as a measure of health outcomes. It includes measures of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ visual analogue scale (VAS) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents.
Change in Quality of Life in Alzheimer's Disease (QOL-AD) | Baseline to Week 12 and Baseline to Week 24
  The QOL-AD is a series of questions designed to be administered to individuals with dementia, to obtain a rating of a patient's quality of life from both the patient and the caregiver. It includes assessments of the individual's relationship with friends and family, concerns about finances, physical condition, mood, and an overall assessment of life quality. There are 13 items with a score range from 13 to 52.
Change in Neuropsychiatric Inventory Questionnaire (NPI) - including Caregiver Distress ratings | Baseline to Week 12 and Baseline to Week 24
  The NPI assesses neuropsychiatric symptoms during routine clinical settings. Namely, the frequency, severity and level of distress caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and appetite/eating disorders).

OTHER OUTCOMES:
Device related Adverse Events | Baseline to Week 12 and Baseline to Week 24
  Device safety assessed according to number of device-related adverse events throughout the course of the study
Rates of epistaxis in aspirin/anti-coagulant users | Baseline to Week 24 compared to 24 weeks prior to study intervention
  The rates of epistaxis in aspirin/anti-coagulant users will be recorded at each study visit and compared to that reported (at baseline) by the subject/caregiver during the prior 24 week period.
Rates of nasal infection | Baseline to Week 24 compared to 24 weeks prior to study intervention
  The rates of nasal infection will be recorded at each study visit and compared to that reported (at baseline) by the subject during the prior 24 week period.
Rates of device/treatment anxiety | Baseline to Week 24
  The rates of device/treatment anxiety as assessed by the Neuropsychiatric Inventory Questionnaire - Anxiety subdomain
Rates of device/treatment anxiety | Baseline to Week 24
  The rates of device/treatment anxiety as assessed by the Zarit Caregiver Burden Interview

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Fischer, MD, Principal Investigator — Unity Health Toronto
Locations (9):
- Headlands Research Orlando, Orlando, Florida, United States
- Canada (8):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Healthtech Connex /Fraser Health, Surrey, British Columbia
  - True North Clinical Research, Halifax, Nova Scotia
  - Bruyère Research Institute, Ottawa, Ontario
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Baycrest, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No